CLINICAL TRIAL: NCT02292615
Title: Application of Integrated MR-PET in Patients With Gynecologic Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201402075MIND
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: MR-PET Imaging
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (3):
- cervical cancer: Group 1: Patients with newly diagnosed gynecologic cancers (including cervical, endometrial, and ovarian cancers).
  Interventions: Other: Medical Imaging
- endometrial cancer: Group 2: Patients with suspicious recurrent gynecologic cancers (including cervical, endometrial, and ovarian cancers).
  Interventions: Other: Medical Imaging
- ovarian cancer: Group 3: Patients with ovarian cancer who had debulking surgery and are going to receive adjuvant chemotherapy.
  Interventions: Other: Medical Imaging

INTERVENTIONS:
Other: Medical Imaging

SUMMARY:
In this prospective cohort study, patients with newly diagnosed gynecologic cancers (including cervical, endometrial, and ovarian cancers) and patients with suspicious recurrent gynecologic cancers will be enrolled. The study period is two years and the estimated patient number is about 220. Patients will undergo image study before and after treatment. The diagnostic accuracy of MR-PET in cancer staging and the potential image biomarkers to monitor treatment response and predict treatment outcome will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1: Patients with newly diagnosed gynecologic cancers (including cervical, endometrial, and ovarian cancers).
2. Group 2: Patients with suspicious recurrent gynecologic cancers (including cervical, endometrial, and ovarian cancers).
3. Group 3: Patients with ovarian cancer who had debulking surgery and are going to receive adjuvant chemotherapy.

Exclusion Criteria:

1. Age <20 or >90 years old
2. Contraindication for MRI:
3. Contraindication for MR contrast medium (Cre > 2.0)
4. History of other malignancy
5. Prior arthroplasty of hip or pelvic bone surgery with metallic fixation (may cause artifacts on MRI)
6. Pregnant or lactating women

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with newly diagnosed gynecologic cancers (including cervical, endometrial, and ovarian cancers) and patients with suspicious recurrent gynecologic cancers will be enrolled. The study period is two years and the estimated patient number is about 220.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The imaging biomarkers determined by MR-PET | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Ting-Fang Shih, MD, Principal Investigator — Department of Medical Imaging, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan